CLINICAL TRIAL: NCT02138695
Title: The Evaluation for Prognostic Factors After Catheter Ablation of Atrial Fibrillation: Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0104
Record Dates: First submitted 2014-04-16; First posted 2014-05-14 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Yonsei AF Cohort: Patients with atrial fibrillation who undergoing catheter ablation of atrial fibrillation

SUMMARY:
1. Purpose of the study

1) To explore clinical recurrence associated clinical factors including age, sex, clinical, electrophysiological, anatomical, imaging, and serologic characteristics.

2) To develop simulation model to predict clinical recurrence and the efficacy of catheter ablation 2. Scientific evidence of the study

1. In atrial fibrillation patients, the maintenance of normal sinus rhythm showed significant reduction of mortality.
2. drug therapy with anti-arrhythmic drug showed many complications and side effect, thus non-drug therapy such as catheter ablation is developed.
3. catheter ablation has been performed for 10years world-wide, and showed superior treatment outcome compared with drug therapy.
4. clinical outcome after catheter ablation is affected not only by age, sex and underlying disease, but also by electrophysiologic, imaging, serologic and electroanatomical remodeling of the heart. However, there are few studies concerning these multifactorial variables.

3. Study population

ELIGIBILITY:
Inclusion Criteria:

* patients who undergoing catheter ablation of atrial fibrillation due to symptomatic, drug refractory atrial fibrillation

Exclusion Criteria:

* patients who do not agree with study inclusion
* permanent AF refractory to electrical cardioversion
* AF with valvular disease ≥ grade 2
* patients with left atrial diameter greater than 60mm
* patients with age less than 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with atrial fibrillation who undergoing catheter ablation in Yonsei Cardiovascular hospital, Yonsei university health system, Seoul, Korea.
Sampling Method: Probability Sample
Enrollment: 3100 (Estimated)
Dates: Start 2014-05; Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Clinical recurrence of atrial fibrillation (AF) after catheter ablation | Participants will be followed for 5 year after catheter ablation
  We defined recurrence of AF as any episode of AF or atrial tachycardia lasting longer than 30 sec. Patients were asked to attend scheduled outpatient follow-up appointments 2, 6, 12, 18, 24, 36, 48 and 60 months after catheter ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho S, Kim D, Park H, Kwon OS, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Pak HN. Mapping and ablation outcomes of extra-pulmonary vein triggers in atrial fibrillation: single-centre retrospective study with consistent provocation protocol. Europace. 2025 Oct 7;27(10):euaf225. doi: 10.1093/europace/euaf225. PMID 40974035
- [Derived] Hwang T, Lim B, Kwon OS, Kim MH, Kim D, Park JW, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Hwang C, Pak HN. Clinical usefulness of digital twin guided virtual amiodarone test in patients with atrial fibrillation ablation. NPJ Digit Med. 2024 Oct 23;7(1):297. doi: 10.1038/s41746-024-01298-z. PMID 39443659
- [Derived] Park JS, Cho I, Kim D, Kim MH, Park JW, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Pak HN. Differentiating Left Atrial Pressure Responses in Paroxysmal and Persistent Atrial Fibrillation: Implications for Diagnosing Heart Failure With Preserved Ejection Fraction and Managing Atrial Fibrillation. J Am Heart Assoc. 2024 Sep 3;13(17):e035246. doi: 10.1161/JAHA.124.035246. Epub 2024 Aug 27. PMID 39189473
- [Derived] Jin Z, Hwang T, Kim D, Lim B, Kwon OS, Kim S, Kim MH, Park JW, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Pak HN. Anti- and pro-fibrillatory effects of pulmonary vein isolation gaps in human atrial fibrillation digital twins. NPJ Digit Med. 2024 Mar 26;7(1):81. doi: 10.1038/s41746-024-01075-y. PMID 38532181
- [Derived] Park YJ, Park JW, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Pak HN. Sex difference in atrial fibrillation recurrence after catheter ablation and antiarrhythmic drugs. Heart. 2023 Mar 10;109(7):519-526. doi: 10.1136/heartjnl-2021-320601. PMID 35332048
- [Derived] Kim M, Yu HT, Kim TH, Lee DI, Uhm JS, Kim YD, Nam HS, Joung B, Lee MH, Heo JH, Pak HN. Ischemic Stroke in Non-Gender-Related CHA2DS2-VA Score 0~1 Is Associated With H2FPEF Score Among the Patients With Atrial Fibrillation. Front Cardiovasc Med. 2022 Feb 8;8:791112. doi: 10.3389/fcvm.2021.791112. eCollection 2021. PMID 35211517
- [Derived] Kwon OS, Hong M, Kim TH, Hwang I, Shim J, Choi EK, Lim HE, Yu HT, Uhm JS, Joung B, Oh S, Lee MH, Kim YH, Pak HN. Genome-wide association study-based prediction of atrial fibrillation using artificial intelligence. Open Heart. 2022 Jan;9(1):e001898. doi: 10.1136/openhrt-2021-001898. PMID 35086918
- [Derived] Kim M, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Pak HN. One-Year Change in the H2FPEF Score After Catheter Ablation of Atrial Fibrillation in Patients With a Normal Left Ventricular Systolic Function. Front Cardiovasc Med. 2021 Aug 3;8:699364. doi: 10.3389/fcvm.2021.699364. eCollection 2021. PMID 34414218
- [Derived] Pak HN, Park JW, Yang SY, Kim M, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH. Sex differences in mapping and rhythm outcomes of a repeat atrial fibrillation ablation. Heart. 2021 Dec;107(23):1862-1867. doi: 10.1136/heartjnl-2020-318282. Epub 2021 Jan 22. PMID 33483352
- [Derived] Park JW, Yu HT, Kim TH, Uhm JS, Joung B, Lee MH, Hwang C, Pak HN. Atrial Fibrillation Catheter Ablation Increases the Left Atrial Pressure. Circ Arrhythm Electrophysiol. 2019 Apr;12(4):e007073. doi: 10.1161/CIRCEP.118.007073. PMID 30917688
- [Derived] Kim TH, Lee JS, Park J, Park JK, Uhm JS, Joung B, Lee MH, Pak HN. Blunted rate-dependent left atrial pressure response during isoproterenol infusion in atrial fibrillation patients with impaired left ventricular diastolic function: a comparison to pacing. Europace. 2015 Oct;17 Suppl 2:ii89-96. doi: 10.1093/europace/euv239. PMID 26842122
- [Derived] Choi EK, Park JH, Lee JY, Nam CM, Hwang MK, Uhm JS, Joung B, Ko YG, Lee MH, Lubitz SA, Ellinor PT, Pak HN. Korean Atrial Fibrillation (AF) Network: Genetic Variants for AF Do Not Predict Ablation Success. J Am Heart Assoc. 2015 Aug 13;4(8):e002046. doi: 10.1161/JAHA.115.002046. PMID 26272656